CLINICAL TRIAL: NCT02266160
Title: EMLA 5% as a Treatment for Tinnitus and Its Accompanied Symptoms
Brief Title: Treating Tinnitus Using Eutectic Mixture of Local Anesthetics (EMLA) 5% Cream
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0055-14
Record Dates: First submitted 2014-09-22; First posted 2014-10-16 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Tinnitus
Keywords: tinnitus; local anaesthetic; EMLA cream 5%
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): 71 tinnitus patients treated with 2 gram EMLA 5% cream a day for 4 days, 4 hours a day.
  we will compare the questionnaires results before and after 4 days of treatment to see whether EMLA cream changes the degree of suffer from tinnitus
  Interventions: Drug: EMLA cream 5%
- 2 (Sham Comparator): 71 tinnitus patients using cetomacrogol cream (lotion cream, does not contain any drug) for 4 days. these patients will fulfill the questionnaires as the investigational group.
  Interventions: Other: cetomacrogol cream (lotion cream)

INTERVENTIONS:
Drug: EMLA cream 5% — the interventional group will spread 2 grams (2 m"l) of EMLA cream over the post auricular area. after 4 hours the patient will wash away the cream. the treatment will last 4 days.
  Other Names: no other names
  Arms: 1
Other: cetomacrogol cream (lotion cream) — lotion cream that does not contain active drug. has no contraindications
  Arms: 2

SUMMARY:
The investigators like to learn whether EMLA cream 5% helps tinnitus patients. so far it is known that lidocaine I.V do helps tinnitus but until now it is not clear if topical anaesthetics (e.g EMLA cream) helps tinnitus.

The investigators are going to compare 4 days of treatment of EMLA 5% cream Versus (VS.) cetomacrogol cream (water- based lotion cream) in treating tinnitus patients.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether EMLA 5% cream decreases tinnitus by comparing pretrial questionnaires to post trial questionnaires.

first we are going to invite tinnitus patients for the first visit. in the first visit we will confirm that the patients is suitable for the trial (no exclusion criteria are present) , perform ear investigation to exclude ear inflammation, perform audiometry to prove sensorineural hearing loss. then the patient will fill 3 questionnaires that reflect the tinnitus severity and show how much the patient does suffer from this conditions. the questionnaires are- beck depression index, tinnitus handicap inventory, Pittsburgh sleep quality index.

Then we will perform randomization: the investigational group will get EMLA 5% cream, the control group will get cetomacrogol cream (a lotion cream).

In the next 4 days the patients (investigational and control groups) will spread the cream for 4 hours a day in the post auricular area of the ear/ ears that suffer/s from tinnitus.

The patient will be instructed to stop the spreading and call the chief investigator When any kind of side effect occurs (topical/ systemic)after 4 days of treatment the patient will come to the clinic once again and fill the same questionnaires. 3 weeks after the beginning of the trial the patient will fill the questionnaires for the third time.

Regarding the questionnaires:

1. Beck depression questionnaire is a 21-questions exam that checks the depression level of the patient. The minimum score is 1 the maximum is 63. The investigators hypotheses states that EMLA cream treatment decreases the Beck questionnaire score
2. Pittsburgh sleep quality index is a 9 questions exam that measure the quality of sleep. the range of results goes between 0-24. The higher the score- the worse is the quality of sleep. The investigators hypotheses states that EMLA treatment improves the results of the Pittsburgh sleep quality questionnaires.
3. Tinnitus handicap inventory estimates the degree that tinnitus affects patients life. it contains 25 questions . The minimum score is 0 and the maximum is 100 . The investigators hypotheses that EMLA cream treatment decreases the score of this questionnaire which means that EMLA cream improves patients quality of life.

ELIGIBILITY:
Inclusion Criteria:

* mature (above 18 years old) patients that suffer tinnitus (unilateral/bilateral) with sensorineural hearing loss

Exclusion Criteria:

* patients that are treated for tinnitus( psychological treatment, hearing aid)
* drugs that affect the CNS
* sensitivity to amide anaesthetic
* hepatic failure
* usage of antiarrhythmic drugs
* severe depression any patients that develops during the trial local/ systemic symptoms such as rash, pain, itching, fever, nervousness,palpitations will be omitted from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
questionnaire results- Beck depression questionnaire | after 4 days of treatment
  Beck depression questionnaire: A 21- questions exam that checks the depression level of the patient. the minimum score is 1 and the maximum score is 63. The investigators hypotheses states that EMLA cream treatment decreases the Beck questionnaire score
questionnaire results- Pittsburgh sleep quality index | after 4 days of treatment
  Pittsburgh sleep quality index : A 9 questions exam that measure the quality of sleep. The range of results goes between 0-24. The higher the score - the worse is the quality of sleep. The investigators hypotheses states that EMLA treatment improves the results of Pittsburgh sleep quality index
questionnaire results- tinnitus handicap inventory | after 4 days of treatment
  tinnitus handicap inventory: estimates the degree that tinnitus affects patients life. It contains 25 questions. The minimum score is 0 and the maximum is 100. The investigators hypotheses that EMLA cream treatment decreases the score of this questionnaire which means that EMLA cream improves patients quality of life

SECONDARY OUTCOMES:
questionnaire results - Beck depression questionnaire | 2 weeks after the beginning of treatment
  estimation of this questionnaire after 2 weeks of treatment
questionnaire results- Pittsburgh sleep quality index | 2 weeks after the beginning of treatment
  estimation of this questionnaire after 2 weeks of treatment
questionnaire results- tinnitus handicap inventory | 2 weeks after the beginning of treatment
  estimation of this questionnaire after 2 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: salim mazzawi, MD, Study Chair — ENT department , "Haemek" hodpital, Afula, ISRAEL

IPD SHARING:
Plan to Share IPD: No